CLINICAL TRIAL: NCT03658434
Title: Palliative Radiotherapy to Dominant Symptomatic Lesion in Patients With Hormone Refractory Prostate Cancer
Acronym: PRADO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRADO
Record Dates: First submitted 2018-07-30; First posted 2018-09-05 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Hormone-refractory Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- feasibilty (Experimental): Palliative Radiotherapy
  Interventions: Radiation: Palliative radiotherapy

INTERVENTIONS:
Radiation: Palliative radiotherapy — Palliative Radiotherapy to Dominant Symptomatic Lesion in Patients With Hormone Refractory Prostate Cancer
  Other Names: PRADO

SUMMARY:
The aim of the present feasibility study of a new short palliative radiotherapy regime that apply to patients with metastatic hormone refractory prostate cancer (HRPC) presenting with a dominating debilitating symptom. Diffusion weighted magnetic resonance imaging (DWI) will apply to identify both the lesion and the most aggressive part of the lesion. The symptomatic lesions will be treated with a dose of 4 x 5 Gy, while for the most aggressive part of the lesion the dose will be escalated to 4 x 7 Gy using a simultaneous integrated boost (SIB) technique.

DETAILED DESCRIPTION:
Please refer to uploaded Study Protocol

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hormone refractory biopsy proven prostate cancer
2. Presenting with a dominating debilitating symptom
3. Expected median survival of 12 months
4. Focal irradiation of lesion is feasible
5. Systemic therapy according to guidelines
6. age ≥18 years
7. Legal capacity, able to understand consequences of the trial
8. Written informed consent

Exclusion Criteria:

1. Relevant comorbidity (limiting radiotherapy according to protocol)
2. Prior radiotherapy limitations to administer radiotherapy according to protocol
3. No large metal implants in vicinity of lesion
4. Department dose constraints for normal tissue can't be met
5. Large bony lesions with extensive osseous destruction
6. Patients symptoms do not correlate with MR findings

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of study participants that complete the study | 6 months
  Proportion of study participants that complete radiotherapy with ≥ 90% of prescribed dose

SECONDARY OUTCOMES:
Response in dominating symptom score (short form McGill pain Questionnaire) | Baseline, 1,3 and 6 months after radiotherapy
  Patient score symptom/pain using the short form McGill pain Questionnaire version 2
Acute radiation toxicity score using CTCAE | Baseline, 1,3 and 6 months after radiotherapy
  Doctor score acute radiation toxicity using the CTCAE version 4
Quality of life score using EORTC QLQ-C30 | Baseline and 6 months after radiotherapy
  Patient fill out EORTC quality of life Questionnaire form C30

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Carl, Phd, Study Chair — Oncology, Zealand University Hospital
Locations (3):
- Dep. Radiation Oncology, Zealand University Hospital, Næstved, Region Sjælland, Denmark
- Germany (2):
  - University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein
  - University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Defined in Partner Agreement Contract
Supporting Information: Study Protocol, SAP
Time Frame: 1. august 2018
Access Criteria: Innocan Partners

REFERENCES:
- [Derived] Carl J, Rades D, Doemer C, Setter C, Dunst J, Hollander NH. Palliative radiotherapy to dominant symptomatic lesion in patients with hormone refractory prostate cancer (PRADO). Radiat Oncol. 2019 Jan 10;14(1):3. doi: 10.1186/s13014-019-1209-0. PMID 30630502

DOCUMENTS (1):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03658434/Prot_000.pdf